CLINICAL TRIAL: NCT06606717
Title: Effects of Resistance-band Training and Nutritional Supplementation in Healthy Older Adults
Brief Title: Effects of Resistance-band Training and Creatine and Whey Protein
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Darren Candow, Professor, University of Regina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 825
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Sarcopenia in Elderly
Keywords: Resistance Exercise; Creatine; Whey Protein; Strength; Lean Mass
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Creatine Whey Protein (Experimental)
  Interventions: Dietary Supplement: Creatine Whey Protein
- Whey Protein (Experimental)
  Interventions: Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Creatine Whey Protein — 3 grams creatine + 30 grams whey protein
  Arms: Creatine Whey Protein
Dietary Supplement: Whey Protein — 30 grams Whey Protein
  Arms: Whey Protein

SUMMARY:
The primary purpose of this research is to compare the effects of creatine monohydrate and/or whey protein supplementation during the first 10 weeks of a 20-week resistance-band training program on measures of body composition (whole-body lean tissue mass, total body water), arm and leg muscle thickness, upper- and lower-body muscle performance (i.e., strength, endurance) and functional ability (walking speed, balance). A secondary purpose of this research is to examine the effects of supplementation cessation (i.e., no creatine and/or whey protein supplementation) during the final 10 weeks of the 20-week resistance-band training program on these measures.

DETAILED DESCRIPTION:
Sarcopenia, characterized by the age-related reduction in strength, muscle mass, and physical function, decreases the ability to perform activities of daily living. Physical inactivity and inadequate nutrition are contributing factors to the development of sarcopenia. Resistance training is a safe, viable and effective intervention which increases measures of muscle and bone mass, muscle performance (i.e., strength, endurance) and functional ability in older adults. However, older adults indicate that high costs and difficulty finding training programming and/or facilities are barriers to participating in resistance training. Home-based resistance-band training is safe, effective and serves as a viable alternative to traditional resistance training (i.e., involving free-weights and machine-based equipment). From a healthy aging perspective, resistance-band training elicits similar improvements in strength (primary indicator of sarcopenia) and functional ability compared to traditional resistance training in older adults. In addition to resistance training (involving resistance-bands), creatine and whey protein supplementations have also been shown to have favorable effects on measures of muscle, bone and functional ability in older adults. However, no study has examined the effects of resistance-band training and creatine and whey protein supplementation in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Untrained (defined as those performing ≤ 1 resistance training session per week for ≥ 6 weeks prior to the start of the study)

Exclusion Criteria:

* Taking creatine monohydrate within 30 days prior to the start of the study
* Currently ingesting whey protein
* Have pre-existing allergies to latex, fruit, dairy, nuts, seafood and mustard

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Whole-body lean mass (kg) | baseline, week 10, week 20
  Bioelectrical impedance analysis
Strength (kg) | baseline, week 10, week 20
  1-repetition maximum leg press and chest press
Endurance (number of repetitions to fatigue) | baseline, week 10, week 20
  Leg press and chest press
Balance (Centre of Pressure) | baseline, week 10, week 20
  Force Plate
Hydration (kg) | baseline, week 10, week 20
  Bioelectrical impedance analysis
Gait Speed (meters) | baseline, week 10, week 20
  Walking distance
Muscle Hypertrophy (cm) | baseline, week 10, week 20
  B-mode ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Darren Candow, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No